CLINICAL TRIAL: NCT01617759
Title: Diagnostic Study on the Performance of an Aspergillus-specific Nested PCR Assay in Cerebrospinal Fluid Samples of Immunocompromised Patients for Detection of Central Nervous System Aspergillosis
Brief Title: Aspergillus-specific PCR Assay in Cerebrospinal Fluid Samples for Detection of Central Nervous System Aspergillosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dieter Buchheidt, Senior Lecturer, Heidelberg University
Other Study IDs: Asp-PCR-CSF
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Aspergillosis; Infection in an Immunocompromised Host
MeSH Terms: conditions — Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — fungal DNA from CSF samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Central nervous system (CNS) invasive aspergillosis (IA) is a fatal complication in immunocompromised patients. Confirming the diagnosis is rarely accomplished as invasive procedures are hampered by neutropenia and low platelet count. Cerebrospinal fluid (CSF) cultures or galactomannan (GM) regularly yield negative results thus suggesting the need for improving diagnostics. Therefore the performance of an established Aspergillus-specific nested PCR in CSF samples of immunocompromised patients with suspicion of CNS IA will be evaluated.

DETAILED DESCRIPTION:
Central nervous system (CNS) invasive aspergillosis (IA) is a fatal complication in immunocompromised patients with hematological malignancies. Confirming the diagnosis is rarely accomplished as invasive procedures are impaired by neutropenia and low platelet count. Cerebrospinal fluid (CSF) cultures or galactomannan (GM) regularly yield negative results thus suggesting the need for improving diagnostic tools. Therefore the performance of an established Aspergillus-specific nested PCR assay in CSF samples of immunocompromised patients with suspicion of CNS IA will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised patients with suspected CNS infection, especially cerebral aspergillosis

Exclusion Criteria:

* proven CNS infections caused by pathogens other than Aspergillus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Immunocompromised individuals
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-09; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Test sensititivity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Buchheidt, MD, Principal Investigator — Mannheim University Hospital, University of Heidelberg, Germany
Locations (1):
- Mannheim University Hospital, Mannheim, Germany